CLINICAL TRIAL: NCT06892665
Title: The Effect Of Using Hypotension Prediction Index To Reduce Intraoperative Hypotension In Caesarean Sections: A Randomised Controlled Trial
Brief Title: The Effect of HPI to Reduce Intraoperative Hypotension in Caesarean Sections
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JEP-2024-463
Record Dates: First submitted 2025-03-09; First posted 2025-03-25 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy Related; Hypotension; Maternal-Fetal Relations; Cesarean Section Complications
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: A prospective, double-blinded, randomised controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: By computer randomisation, patients will be randomised into two groups, Group A (Intervention: HPI) or Group B (control: oNIBP). Standard monitoring will be applied, including a 3-lead electrocardiogram, pulse oximetry, and oNIBP in the upper arm. The oNIBP monitoring will be performed every 1 minute before, and every 3 minutes after the baby is delivered, up to 90 minutes of surgery duration. After 90 minutes, data collection will cease. In addition to the standard monitoring, all patients will have an Acumen IQ cuff placed on one of their fingers, as Appendix A shows, connected to haemodynamic monitoring using HemoSphere (Edwards Lifesciences) with HPI software enabled. In Group A, the Acumen IQ cuff, with HPI and other haemodynamics parameters, is available to the anaesthetist to view and act upon. While in Group B, the attending anaesthetist will be blinded from the HPI parameters.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: HPI Group (Experimental): There were 2 arm group, in Group 1the Acumen IQ cuff, with HPI and other haemodynamics parameters, is available to the anaesthetist to view and act upon.
  Interventions: Device: Hypotension prediction index
- Group 2: NIBP Group (Placebo Comparator): the attending anaesthetist will be blinded from the HPI parameters.
  Interventions: Device: Non invasive Blood Pressure Monitoring

INTERVENTIONS:
Device: Hypotension prediction index — HPI and other haemodynamics parameters, is available to the anaesthetist to view and act upon
  Other Names: HPI
  Arms: Group 1: HPI Group
Device: Non invasive Blood Pressure Monitoring — Anaesthetist will respond to hemodynamic variables using NIBP
  Other Names: NIBP
  Arms: Group 2: NIBP Group

SUMMARY:
During caesarean section, blood pressure variations especially a reduction in blood pressure (or hypotension) can bring harmful effects to mother and baby. This usually occurs after spinal anaesthesia is administered. Usually, the anaesthetist will treat hypotension as it occurs. However, a new medical device is now available to predict hypotension. It is called the Hypotension Prediction Index (HPI). This device allows the prediction of hypotension; hence, treatment can be given before it occurs. It has been widely utilised in major surgeries like abdominal tumour surgery and cardiac surgery worldwide and has shown a substantial reduction in hypotension. This study aims to determine whether the duration and severity of hypotension can be reduced when HPI is used in lower segment caesarean sections. The secondary objective of the study is to determine if the complication rate can be reduced in both mother and baby.

DETAILED DESCRIPTION:
Hypotension Prediction Index (HPI) has been shown to reduce IOH significantly in non-cardiac and major abdominal surgeries.The role of HPI beyond reducing IOH has also been a subject of research. Andrzejeska et al. demonstrated that the use of HPI in adolescent idiopathic scoliosis surgery leads to lower reductions in post-surgery haemoglobin levels, shorter duration of hypotension and shorter hospital admissions. Additionally, the intervention group had shorter timeframes from the end of surgery to extubation.

The development of a non-invasive finger blood pressure device compatible with HPI called the Acumen IQ cuff, made it possible to use HPI without inserting an arterial catheter. The arterial pressure waveform generated by a non-invasive finger cuff was reliable and in agreement with the radial artery blood pressure. A retrospective analysis was conducted by Frassanito et al. to determine the performance of HPI using arterial waveform recorded by a non-invasive finger probe to predict hypotension in patients undergoing CS under spinal anaesthesia. They have found that HPI, using this non-invasive probe, was able to predict hypotension with a sensitivity and specificity of 83% and 83% at 3 minutes, 97% and 97% at 2 minutes, and 100% and 100% at 1 minute, before it occurs.

This study aims to determine if the solution to reduce IOH lies in predicting intraoperative hypotension during lower segment ceaserean section (CS). The benefits of HPI may extend beyond reducing the incidence and severity of IOH, to bringing positive outcomes to the foetus. This study will determine whether integrating an early warning system produces benefits significant enough to justify changing our anaesthetic practice.

PROBLEM STATEMENT

Varying methods have been utilised to reduce IOH in CS. A novel software, HPI, was developed to predict hypotension, enabling clinicians to institute guided treatment before maternal hypotension occurs. The investigator need to determine if HPI has benefits in CS, thus leading to better maternal and neonatal outcomes.

RESEARCH QUESTION

Can HPI using the non-invasive continuous arterial pressure waveforms reduce the duration and severity of hypotension in patients undergoing CS under spinal anaesthesia?

OBJECTIVES

Study objective:

To determine if HPI has benefits in CS, thus leading to better maternal and neonatal outcomes compared to oNIBP.

Primary outcome:

The duration and severity of hypotensive events reported as a time-weighted average (TWA) - MAP < 65 mmHg in HPI group (intervention) versus standard oNIBP.

Secondary outcomes:

1. To determine whether the use of HPI leads to better maternal outcomes (incidence of nausea and vomiting, blood loss, length of hospital stay, maternal satisfaction, incidence of surgical site infection)
2. To determine whether the use of HPI leads to better foetal outcomes (Apgar scores, umbilical cord pH, length of hospital stay)
3. To determine the amount of vasopressors and inotropes administered throughout CS if HPI is used versus conventional oNIBP monitoring

RESEARCH HYPOTHESIS

Additional parameters from HPI in the CS under spinal anaesthesia will reduce the duration and severity of intraoperative hypotension and provide better maternal and neonatal outcomes.

ELIGIBILITY:
Inclusion criteria:

* ≥ 37 weeks of gestation
* Elective CS
* Age between 18 - 40 years old
* Singleton pregnancy
* Planned for spinal anaesthesia

Exclusion criteria:

* American Society of Anesthesiologists (ASA) III and above
* Body mass index (BMI) ≥ 40 kg/m2
* Increased risk of developing peripartum haemorrhage
* History of peripartum haemorrhage
* Placenta previa major, accrete, increta, percreta
* Gravida ≥ 5
* Presence of large uterine fibroids
* Congenital bleeding disorders such as Haemophilia A, Haemophilia B and Von Willebrand disease
* Acquired bleeding disorders such as thrombocytopenia and coagulopathy
* Contraindications to finger cuff orNIBP application, such as finger ischaemia, upper limb neurological deficit, discoloured nail
* Cardiac arrhythmias and aortic regurgitation
* Patient's refusal

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Parturients
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Time-weighted average of Mean arterial pressure <65mmHg | From spinal anaesthesia to completion of surgery
  Calculated using a formula. TWA-MAP < 65 mmHg = (the depth of hypotension< MAP of 65 mmHg x time spent below a MAP of 65 mmHg (minutes))/(total duration of operation (minutes))

SECONDARY OUTCOMES:
Incidence of nausea and vomiting, | Perioperative up to 2 days
  Maternal incidence of nausea and vomiting
length of hospital stay | Perioperative up to 2 weeks
  maternal length of hospital stay
maternal satisfaction | Perioperative up to 2 weeks
  Likert scale from 1 (very unsatisfied) to 5 (very satisfied)
incidence of surgical site infection | Perioperative up to 2 weeks
  maternal surgical site infection
Apgar score of feotal | 1 minute and 5 minutes after delivery
  Apgar scores of 0-10 ( Apgar score of 7 and more is considered normal)
Umbilical cord PH | Immediately upon delivery of baby
  Umbilical cord PH taken after after delivery of baby
Neonatal length of stay | Perioperative up to 2 weeks
  Neonatal length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Azlina Masdar, Principal Investigator — National University of Malaysia
Locations (1):
- Hospital Canselor Tuanku Muhriz, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
The data of the study will be available in public data repository
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After completion of the study and analysis for 5 years
Access Criteria: With permission from corresponding author

REFERENCES:
- [Background] Murabito P, Astuto M, Sanfilippo F, La Via L, Vasile F, Basile F, Cappellani A, Longhitano L, Distefano A, Li Volti G. Proactive Management of Intraoperative Hypotension Reduces Biomarkers of Organ Injury and Oxidative Stress during Elective Non-Cardiac Surgery: A Pilot Randomized Controlled Trial. J Clin Med. 2022 Jan 13;11(2):392. doi: 10.3390/jcm11020392. PMID 35054083
- [Background] Sun LY, Wijeysundera DN, Tait GA, Beattie WS. Association of intraoperative hypotension with acute kidney injury after elective noncardiac surgery. Anesthesiology. 2015 Sep;123(3):515-23. doi: 10.1097/ALN.0000000000000765. PMID 26181335
- [Background] Frassanito L, Sonnino C, Piersanti A, Zanfini BA, Catarci S, Giuri PP, Scorzoni M, Gonnella GL, Antonelli M, Draisci G. Performance of the Hypotension Prediction Index With Noninvasive Arterial Pressure Waveforms in Awake Cesarean Delivery Patients Under Spinal Anesthesia. Anesth Analg. 2022 Mar 1;134(3):633-643. doi: 10.1213/ANE.0000000000005754. PMID 34591796
- [Background] Andrzejewska A, Miegon J, Zacha S, Skonieczna-Zydecka K, Jarosz K, Zacha W, Biernawska J. The Impact of Intraoperative Haemodynamic Monitoring, Prediction of Hypotension and Goal-Directed Therapy on the Outcomes of Patients Treated with Posterior Fusion Due to Adolescent Idiopathic Scoliosis. J Clin Med. 2023 Jul 9;12(14):4571. doi: 10.3390/jcm12144571. PMID 37510686